CLINICAL TRIAL: NCT01869881
Title: Effect of Sarpogrelate On the Nephropathy in Type 2 Diabetes
Brief Title: Effect of Sarpogrelate On the Nephropathy in Type 2 Diabetes (SONATA Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YCM009
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sarpogrelate (Active Comparator)
  Interventions: Drug: Anplag(Sarpogrelate)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anplag(Sarpogrelate) — Sarpogrelate 100mg 2 tablets, bid, 400mg/day
  Arms: Sarpogrelate
Drug: Placebo — Placebo 100mg 2 tablets, bid, 400mg/day
  Arms: Placebo

SUMMARY:
Phase 4 Study to evaluate the safety and effect on decreasing subjects' albuminuria who have Type 2 Diabetes by using sarpogrelate and placebo.

ELIGIBILITY:
Inclusion Criteria:

* person who signed on ICF
* Type 2 diabetic patient who have microalbuminuria or overt proteinuria
* In case of hypertension patients, who keep the same medication steadily over last 4 weeks

Exclusion Criteria:

* patients who have hypersensitivity on sarpogrelate or other salicylic acid
* patients who should keep the antiplatelet agent because of acute cardiac disease or peripheral vein disease
* patients who took other anticoagulant agent within 1 month
* patient who take ACEI OR ARB but not controlled(over 150/100mmHg)
* Type 1 diabetes patients
* Patient who have cardiac or liver problem
* Cr: >1.8mg/dl or GFR: <40ml/min
* malignant tumor patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-11-17 (Actual); Study Completion 2015-01-28 (Actual)

PRIMARY OUTCOMES:
ACR(Urine Albumin/Creatinine ratio) | treatment period(24 weeks)
  change of percentage

SECONDARY OUTCOMES:
ACR(Urine Albumin/Creatinine ratio) | Treatment period(24 weeks)
  improvement efficiency rate of ACR comparing to baseline Definition of improvement efficiency : ACR become normal(<20mg/g Cr) or ACR is decreased more than 50% comparing to data before taking IP(Investigators' product)
urinary 5-HIAA(5-Hydroxyindoleacetic acid), type 4 collagen | treatment period(24 weeks)
  changes comparing to baseline data
ACR(Urine Albumin/Creatinine ratio) | treatment period(24 weeks)
  improved amount comparing to baseline data
ACR(Urine Albumin/Creatinine ratio) | treatment period(24 weeks)
  rate of normalized ACR
Creatinine | treatment period(24 weeks)
  improved amount of Creatinine
PCR(Protein to Creatinine ratio in Urine) | treatment period(24 weeks)
  improved rate comparing to baseline data

CONTACTS AND LOCATIONS:
Overall Officials: D.S Choi, MD, PhD, Principal Investigator — Korea University Hospital, Anam
Locations (1):
- Korea University, Anam, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730